CLINICAL TRIAL: NCT00886704
Title: Influence of Dietary Omega-3 Fatty Acids in a Convenience Drink (Smartfish) on the Omega-3 Index in Patients With Atherosclerotic Disease
Brief Title: Omega-3 Fatty Acids, the Omega-3 Index, and Atherosclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Clemens von Schacky, Preventive Cardiology, University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 477-08
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2009-07

CONDITIONS: Atherosclerosis
Keywords: Omega-3 fatty acids; dietary supplementation; atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Convenience drink with EPA and DHA (Active Comparator): Daily consumption of 200 ml convenience drink, containing 0.5 g EPA and DHA (Omega-3 Fatty Acids)
  Interventions: Dietary Supplement: 500 mg eicosapentaenoic (EPA) plus docosahexaenoic acids (DHA)
- Convenience drink without EPA and DHA (Placebo Comparator): Daily consumption of 200 ml convenience drink, not containing 0.5 g EPA and DHA (Omega-3 Fatty Acids), but containing 1.0 g of Omega-6 Fatty Acids (e.g. corn oil)
  Interventions: Dietary Supplement: 500 mg eicosapentaenoic (EPA) plus docosahexaenoic acids (DHA); Dietary Supplement: Control convenience drink

INTERVENTIONS:
Dietary Supplement: 500 mg eicosapentaenoic (EPA) plus docosahexaenoic acids (DHA) — Composition of active convenience drink (smartfish): 200 ml drink, enriched with 940 mg omega-3 fatty acids, of which 200 mg are EPA, 300 mg DHA and 100 mg DPA, slightly carbonized..
  Energy content 486 kJ (116 kcal), protein 0.6 g, Carbohydrates 22 g, total fat 4 g, of which 0.6 g saturated fatty acids, 1.8 g monounsaturates, 1.4 g polyunsaturates. Vitamin D 0.85 ug.
  Control convenience drink: as above, containing about 1 g Omega-6 fatty acids from e.g. corn oil.
Dietary Supplement: Control convenience drink — Control convenience drink: as above, containing about 1 g Omega-6 fatty acids from e.g. corn oil.
  Arms: Convenience drink without EPA and DHA

SUMMARY:
An increase in intake of omega-3 fatty acids should increase the Omega-3 Index. Current evidence indicates that this may lead to a reduction in risk for sudden cardiac death and atherosclerotic diseases like myocardial infarction. The aim of the study is to investigate, how supplementing a convenience drink with omega-3 fatty acids influences the Omega-3 Index, as compared to an unsupplemented matching convenience drink. Palatability and safety of the drink are also to be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet the current guideline criteria for atherosclerosis, like coronary, peripheral or carotid artery disease, like previous myocardial infarction or acute coronary syndrome, coronary revascularization (operation or transluminally), or positive angiography or ultrasound.
2. Age: 30 - 75 years
3. Low Omega-3 Index (<5%)
4. Subjects must have adequate fluency in German or English to complete baseline and follow-up interviews.
5. Stable intake of food containing EPA+DHA before and during study
6. Subjects must be able and willing to give written informed consent, and to comply with study procedures.

Exclusion Criteria:

1. Subjects for whom the intake of omega-3 fatty acids is mandatory according to recent treatment guidelines or who take omega-3 fatty acids supplements on a regular basis.
2. Patients consuming >2 portions of fatty fish / week
3. Patients with serious bleeding disorder. Use of platelet inhibitors or anticoagulation with a target INR of 2.0 - 3.0 is not an exclusion criterion.
4. Subjects with any acute and life-threatening condition, such as collapse and shock, acute myocardial infarction (last three months), stroke, embolism.
5. Subjects with significant medical co-morbidity, seriously limiting life expectancy or insulin-treated diabetes mellitis or a BMI>30
6. Allergy/intolerance or history of hypersensitivity to components of study intervention, like lactose.
7. Pregnant subjects - due to any possible teratogenic effects of study nutrition on the fetus - and breastfeeding subjects. In addition, women of childbearing potential who will not practice a medically accepted method of contraception will be excluded.
8. Subjects who, in the investigator's judgement, will not likely be able to comply with the study protocol or with known drug- or alcohol abuse/dependence in the past 2 years.
9. Use of any investigational agents within 30 days prior to t0

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clemens von Schacky, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Preventive Cardiology, Munich, Germany

REFERENCES:
- [Result] Kohler A, Bittner D, Low A, von Schacky C. Effects of a convenience drink fortified with n-3 fatty acids on the n-3 index. Br J Nutr. 2010 Sep;104(5):729-36. doi: 10.1017/S0007114510001054. Epub 2010 Apr 27. PMID 20420756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 190 subjects were screened and gave informed consent, and 50 were enrolled.
Pre-assignment Details: The main reason for screen failure (about 95 %) was an omega-3 index < 5.0%. Additional subjects were excluded because of the lack of any evidence for atherosclerotic disease, hospitalisation or lactose intolerance.
Period: Overall Study
Arm/Group | Convenience Drink With EPA and DHA (Omega-3 Fatty Acids) | Convenience Drink Without EPA and DHA
Started | 40 | 10
Completed | 40 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convenience Drink With EPA and DHA (Omega-3 Fatty Acids) | Convenience Drink Without EPA and DHA | Total
Number analyzed (Participants) | 40 | 10 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 5 | 20
  >=65 years | 25 | 5 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 65.1 (6.1) | 64.5 (5.9) | 64.8 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 29 | 5 | 34
Region of Enrollment [Number; unit: participants]
  Germany | 40 | 10 | 50

OUTCOME MEASURES:

1. Secondary Outcome: Palatability
Description: Palatability assessed as number on a visual analogue scale from 0 - 10, with 0 being the worst and 10 being the best possible outcome
Time Frame: at 8 weeks
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: Number on a scale from 0 - 10
Groups:
- Convenience Drink With EPA and DHA; Convenience Drink Without EPA and DHA: Palatability
Arm/Group | Convenience Drink With EPA and DHA | Convenience Drink Without EPA and DHA
Number analyzed (Participants) | 40 | 10
Number on a scale from 0 - 10 | 8.50 (1.84) | 8.39 (1.71)

2. Primary Outcome: Omega-3 Index
Description: Percentage of eicosapentaenoic and docosahexaenoic acids in total red cell fatty acids, as determined with a standardized analytical procedure, i.e. the HS-Omega-3 Index. Currently, the target range for the HS-Omega-3 Index has been suggested to be between 8% and 11%. Cardiovascular risk increases at levels below 8%, whereas levels above 11% do not seem to confer further benefit. Values of the HS-Omega-3 Index have been found between 1.5% and 20%.
Time Frame: after eight weeks of intervention
Measure: Median (Standard Deviation); unit: % EPA+DHA in total red cell fatty acids
Arm/Group | Convenience Drink With EPA and DHA (Omega-3 Fatty Acids) | Convenience Drink Without EPA and DHA
Number analyzed (Participants) | 40 | 10
% EPA+DHA in total red cell fatty acids | 4.37 (0.51) | 4.71 (0.73)

ADVERSE EVENTS:
Arm/Group | Convenience Drink With EPA and DHA (Omega-3 Fatty Acids) | Convenience Drink Without EPA and DHA
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/10
Other Adverse Events (participants affected / at risk) | 0/40 | 0/10

LIMITATIONS AND CAVEATS:
Single center study, too small to detect rare side effects, 8 week intervention period relatively short.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No